CLINICAL TRIAL: NCT01822535
Title: Core Temperature During Cold Exposure in Persons With Tetraplegia
Brief Title: Body Temperature in Persons With Tetraplegia When Exposed to Cold
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, John Handrakis, PT, DPT, EdD, Research Health Science Specialist, James J. Peters Veterans Affairs Medical Center
Allocation: Non-Randomized | Model: Factorial | Masking: None
Other Study IDs: 01374
Record Dates: First submitted 2013-03-21; First posted 2013-04-02 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-02

CONDITIONS: Tetraplegia; Hypothermia; Mild Cognitive Impairment
Keywords: Quadriplegia; Spinal Cord Injuries; Body Temperature Regulation; Mild Cognitive Impairment
MeSH Terms: conditions — Quadriplegia; Hypothermia; Cognitive Dysfunction; Spinal Cord Injuries | interventions — Midodrine; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No Drug: Tetraplegia (No Intervention): Tetraplegia: Lesion level T1 and above, American Spinal Injury Association (ASIA) impairment levels A and B, ages 18-68 years.
  Exposure of up to 2 hours in a cool room.
- No Drug: AB Controls (No Intervention): AB Controls: Matched for age and gender to subjects with tetraplegia. Exposure of up to 2 hours in a cool room.
- Drug (midodrine): Tetraplegia (Experimental): Persons with tetraplegia who completed Visit 1 (no drug). Participants are administered midodrine hydrochloride (10 mg tablet) by a physician before exposure of up to 2 hours in a cool room. (Visit 2)
  Interventions: Drug: Midodrine hydrochloride

INTERVENTIONS:
Drug: Midodrine hydrochloride — Midodrine hydrochloride is an approved medication used to treat low blood pressure. We are using a standard dose of 10 mg (tablet) only one time to determine if the effects of this drug improve the ability to maintain body core temperature in a cool environment (off-label use). A physician will administer the drug once before the cool thermal challenge in subjects with tetraplegia only(Visit 2)
  Other Names: Midodrine hydrochloride 10 mg tablet; Amatine; ProAmatine; Gutron
  Arms: Drug (midodrine): Tetraplegia

SUMMARY:
The ability to maintain normal body core temperature (Tcore = 98.6°F) is impaired in persons with tetraplegia. Despite the known challenges to the ability of persons with spinal cord injury (SCI) to maintain Tcore, and the effects of hypothermia to impair mental function in able-bodied (AB) persons, there has been no work to date addressing these issues in persons with tetraplegia.

The aim of this study is to determine if exposure of up to 2 hrs to cool temperatures (64°F) causes body core temperature to decrease in persons with tetraplegia and if that decrease is related to a decrease in mental performance.

After sitting in a cool (64°F) room for up to 2 hours the investigators hypotheses are:

Hypotheses (1): Tcore of most of the persons with tetraplegia will decline approximately 1.8°F (e.g., 98.6 to 96.8°F) while Tcore of controls will not decline at all; (2) Most of the persons with tetraplegia will show a decline in mental performance (memory or clear-headedness) while only some of AB controls will show a decline.

The second aim of this study is to determine if a 10 mg dose of an approved blood pressure raising medicine (midodrine hydrochloride) will (1) reduce the decrease in body core temperature and (2) prevent or delay the decline in mental performance in the group with tetraplegia compared to the exact same procedures performed on the day with no medicine (Visit 1) in the same group.

Hypotheses (3 & 4): The changes in blood flow to the skin caused by taking a one-time dose of midodrine will lessen the decline in Tcore and prevent or delay the decline in mental performance compared to the changes in Tcore and mental performance during cool temperature exposure without midodrine in the group with tetraplegia.

DETAILED DESCRIPTION:
This study will investigate the mechanisms contributing to the thermoregulatory fragility in persons with tetraplegia when exposed to cool ambient temperatures that are routinely encountered during activities of daily living (ADL). Subnormal body core temperatures and vulnerability to hypothermia (Tcore<95°F) has been reported in veterans with tetraplegia upon exposure to relatively mild environmental temperatures. The impact that a drift in Tcore will be expected to have on cognitive performance, specifically working memory and executive function, will be demonstrated. These 2 areas of cognitive performance are vital for the ability to optimally care for one's self, which persons with higher cord lesions must excel at to ensure health, as well as to be able to attain the maximal degree of independence possible. Administration of an alpha agonist, midodrine hydrochloride, in an attempt to attenuate the drift in Tcore and prevent or delay the expected decline in cognitive performance to exposure to cool on cognitive function will be investigated as well.

Primary Specific Aim: To determine the change in: (1) Tcore and (2) cognitive performance (attention, working memory, processing speed, and executive function) in persons with tetraplegia after exposure to a cool environment (64°F) for up to 120 min in the seated position.

Primary Hypotheses:(1) 66% of persons with tetraplegia will demonstrate a decline of 1.8°F in Tcore while 0% of controls will demonstrate that same thermal decline; (2) 80% of persons with tetraplegia will have a decline of at least 1 T-score in Stroop Interference scores (executive functioning) while 30% of controls will demonstrate that same magnitude of decline.

Secondary Specific Aims: To determine the change in: (1) the average of distal skin temperatures, (2) metabolic rate, and (3) subjective rating of thermal sensitivity after exposure to 64°F in the seated position.

Secondary Hypotheses: Persons with tetraplegia will have less of a percent change in average distal skin temperatures and metabolic rate, and report lower thermal sensitivity ratings compared with AB.

Tertiary Specific Aim: To determine if a single, 10 mg dose of midodrine will (1) reduce the decrease in Tcore and (2) prevent or delay the decline in cognitive performance in the group with tetraplegia.

Tertiary Hypotheses: Because administration of a peripheral alpha-agonist will address the primary thermoregulatory impairment to cool temperature exposure in persons with tetraplegia-that is, lack of vasoconstriction, the midodrine-induced peripheral vasoconstriction will be anticipated to blunt the decrease in Tcore and prevent or delay the decline in cognitive performance compared to cool exposure without drug administration.

Preparation for Study Visits: The study visits will be separated by a minimum of 1 day and no more than 14 days. Subjects will wear minimal clothing (gym shorts, sports bra) during the study to maximize bare skin exposure to the cool temperature. Each subject will be asked to eat a light, standard meal 2 hours prior to their scheduled visit consisting of either a plain bagel or 2 pieces of toast. For each visit they will be asked to empty their bladders prior to arrival and again upon arrival, if needed.

Visit 1: Cold Ambient Challenge: Instrumentation: During Visit 1, all subjects will be transferred to a padded table for instrumentation, after which they will be transferred back to their own wheelchair or, for controls, to a provided wheelchair. All subjects will use a Roho seat cushion for air circulation consistency and decubiti prevention. A rectal probe will be placed 4 inches beyond the anal sphincter for core temperature measurement, and skin thermal sensors will be taped at 15 sites above and below the level of lesion for collection of skin temperatures. A mask will be placed over the subject's nose and mouth for measurement of exhaled gases from which resting metabolic rate will be calculated from analysis of expired gases (VO2) by a metabolic cart. Laser Doppler flowmetry (LDF) will be used to measure changes in microvascular perfusion by taping a doppler probe on the skin in the area of the ulnar styloid processes and medial malleoli bilaterally (wrists and ankles) to confirm vasoconstriction. A pulse oximeter will be placed on the left second digit to obtain blood oxygen saturation and heart rate (HR). An automated blood pressure cuff will be placed above the right elbow to measure brachial BP. An intravenous catheter will be placed in the right antecubital or nearby vein and secured for sequential blood collection for cortisol and norepinephrine.

Baseline Collection: At the end of the 30 minute acclimation period (81°F), a baseline (BL) collection of the following parameters will be performed for 15 minutes with Tcore, skin temperatures, and VO2 measured continuously; HR, BP, blood oxygen saturation, subjective measures of thermal sensitivity, and 5 minutes of LDF will be measured at 10 minute intervals. A venous blood draw will be collected once at baseline for norepinephrine and cortisol concentrations. At the end of the BL period, a cognitive performance battery will be administered.

Thermal Challenge: Following completion of the baseline period, subjects will be wheeled into an 18°C thermal chamber for 120 minutes or until Tcore ≤ 95°F. Tcore, skin temperatures, and VO2 will be continuously monitored to ensure subject safety throughout the protocol; brachial BP, HR, blood oxygen saturation, thermal sensitivity, and symptoms of hypothermia and autonomic dysreflexia will be assessed at 10 min intervals while LDF will be measured for 5 minutes every 20 minutes. Venous blood will be collected at 50 minute intervals. A decrease in Tcore to ≤ 95°F, or moderate subject discomfort, will result in termination of the protocol. The cognitive performance battery will be administered when Tcore has declined 1.8°F or is ≤ 95.9°F (in subjects with tetraplegia) or after 120 minutes of cold exposure (in both groups) on Visits 1 & 2.

Visit 2: Cold Ambient Challenge with Midodrine: Visit 2 will be completed in subjects with tetraplegia who participated in Visit 1 and who had an impaired ability to maintain Tcore. Following completion of the BL period, subjects will be orally administered midodrine hydrochloride (10 mg tablet). Forty minutes after midodrine administration (for onset of drug effect), a second BL collection will be obtained, and subjects will be wheeled into the 64°F thermal chamber for 120 minutes or until Tcore ≤ 95°F. Data collection will follow the same schedule and be conducted in the seated position as in Visit 1. If brachial BP increases to 160/90 mmHg, the subject will be removed from the cool room and evaluated by Dr. William A. Bauman, who may consider the administration of labetalol (to lower BP), if deemed necessary.

ELIGIBILITY:
Inclusion Criteria:

* (1) Between 18 and 68 years of age;
* (2) Duration of injury ≥ 1 year; (2) Level of SCI C3-T1;
* (3) Euhydration (subjects will be instructed to avoid caffeine and alcohol, maintain normal salt and water intake, and avoid strenuous exercise for 24 hours prior to study)

Exclusion Criteria:

* (1) Known coronary heart, kidney, peripheral vascular or cerebral vascular disease;
* (2) High blood pressure;
* (3) Untreated thyroid disease;
* (4) Diabetes mellitus;
* (5) Acute illness or infection;
* (6) Dehydration;
* (7) Known allergies to midodrine hydrochloride;
* (8) Smoking;
* (9) Pregnancy

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Handrakis, PT, DPT, EdD, Principal Investigator — James J Peters VA MC
Locations (1):
- Center of Excellence for the Medical Consequences of SCI, JJP VAMC, 7A-13, The Bronx, New York, United States

REFERENCES:
- [Derived] Handrakis JP, Liu SA, Rosado-Rivera D, Krajewski M, Spungen AM, Bang C, Swonger K, Bauman WA. Effect of Mild Cold Exposure on Cognition in Persons with Tetraplegia. J Neurotrauma. 2015 Aug 1;32(15):1168-75. doi: 10.1089/neu.2014.3719. Epub 2015 Mar 31. PMID 25531297
- See also: Link to Center of Excellence Research Center. Look under Research to find Thermoregulation — http://scirc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Tetraplegia: Lesion level C3-T1, American Spinal Injury Association (ASIA) impairment levels A and B, ages 18-68 years
- Able-bodied (AB): Age- and gender-matched to individuals with tetraplegia.
Period: Visit 1 - Tetraplegia and Able-Bodied
Arm/Group | Tetraplegia | Able-bodied (AB)
Started | 17 | 13
Completed | 11 | 11
Not Completed | 6 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 4 | 2
Period: Visit 2 - Tetraplegia Only - Drug
Arm/Group | Tetraplegia | Able-bodied (AB)
Started | 11 (These subjects were individuals who completed Visit 1 of testing.) | 0 (Able-bodied subjects were not enrolled for a second visit.)
Completed | 10 | 0
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tetraplegia: Lesion level T1 and above, ASIA levels A and B, ages 18-68 years
- Able-bodied: Age- and gender-matched to individuals with tetraplegia.
- Total: Total of all reporting groups
Arm/Group | Tetraplegia | Able-bodied | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 11 | 11 | 22
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Visit 1: Percent Change in Core Body Temperature
Description: We will test the effects of cool temperature (64°F) exposure, of up to 120 minutes, on the ability to maintain a constant body temperature (e.g., core temperature of 98.6°F) in persons with tetraplegia through comparing the percent changes in core body temperatures between groups from baseline to after cool exposure.
Time Frame: Baseline, Up to 2 hours
Population: Only the subjects with tetraplegia who demonstrated sympathetic interruption (insignificant decreases in distal skin temperatures, distal microvascular blood flow (LDF) and decreases of 1.0°C or greater in Tcore during cool exposure), and their matched able-bodied controls were analyzed.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Tetraplegia | Able-bodied
Number analyzed (Participants) | 7 | 7
Percent Change | -1.2 (0.33) | 0.05 (0.21)
Statistical Analysis 1: Comparison: Tetraplegia vs Able-bodied; Between-group differences in percent changes in core body temperature from baseline values to after cool exposure were analyzed. Because individuals with tetraplegia have impaired thermoregulatory mechanisms, we hypothesized that their percent change in core body temperature would be significantly larger than that of able-bodied controls; Test type: Superiority or Other; p < 0.01, ANOVA

2. Secondary Outcome: Visit 1: Percent Changes in Cognitive Performance - Stroop Interference
Description: Cognitive performance will be evaluated using the Interference T-Scores obtained using the Stroop Color and Word Test. We will measure the change in cognitive performance in persons with tetraplegia after exposure to a cool environment (64°F) of up to 120 min in the seated position. Note: Interference T-Scores are derived from the difference between the raw Color-Word score and the projected Color-Word score (which is, in turn, based on the raw scores obtained in the Word and Color portions of the Test). Lower scores indicate poorer performance, and a positive percent change in T-scores indicates improved performance.
Time Frame: Baseline, Up to 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Groups:
- Tetraplegia: Lesion level C3-T1, ASIA levels A and B, ages 18-68 years
Arm/Group | Tetraplegia | Able-bodied
Number analyzed (Participants) | 7 | 7
Percent Change | -3.9 (3.8) | 5.4 (9.2)
Statistical Analysis 1: Comparison: Tetraplegia vs Able-bodied; Between-group comparisons of percent changes in Stroop Interference T-scores from baseline values to after cool exposure were analyzed. We hypothesized that subjects with tetraplegia would have greater declines in cognitive performance after cool exposure than able-bodied controls; Test type: Superiority or Other; p = 0.018, ANOVA

3. Secondary Outcome: Visit 1: Percent Changes in Cognitive Performance - Delayed Recall
Description: Cognitive performance will be evaluated using the Delayed Recall obtained using the Memory section of the Montreal Cognitive Assessment (MoCA). We will measure the change in cognitive performance in persons with tetraplegia after exposure to a cool environment (64°F) of up to 120 min in the seated position. Note: Scores are based on individual performance. All subjects are asked to remember two lists of five words (one list during baseline, and one list during cool Challenge). Lower scores indicate poorer performance, and a positive percent change in indicates improved cognitive performance.
Time Frame: Baseline, Up to 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Tetraplegia | Able-bodied (AB)
Number analyzed (Participants) | 7 | 7
Percent Change | -55.2 (47.4) | 6.4 (49.7)
Statistical Analysis 1: Comparison: Tetraplegia vs Able-bodied (AB); Between-group comparisons of percent changes in Delayed Recall from baseline values to after cool exposure were analyzed. We hypothesized that subjects with tetraplegia would have greater declines in cognitive performance after cool exposure than able-bodied controls; Test type: Superiority or Other; p = 0.0431, ANOVA

4. Primary Outcome: Visit 2: Percent Change in Core Body Temperature With Midodrine
Description: We will test the effects of midodrine on the ability to maintain a constant body temperature (e.g., core temperature of 98.6°F) after exposure to cool temperatures (64°F) in persons with tetraplegia through comparing the percent changes in core body temperature during visit 1 to percent changes in core body temperature during visit 2.
Time Frame: Baseline, Baseline Post-midodrine, Up to 2 hours
Population: Subjects analyzed were individuals who completed visit 1 of testing.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Tetraplegia
Number analyzed (Participants) | 7
Percent Change | -2.2 (0.9)
Statistical Analysis 1: Comparison: Tetraplegia; We hypothesized that administration of midodrine would attenuate the fall in core body temperature. Within-group percent changes in core body temperature were analyzed to compare data from visit 1 (no drug) to visit 2 (drug); Test type: Superiority or Other; p = 0.30, ANOVA

ADVERSE EVENTS:
Time Frame: Throughout the entire study, i.e. 2011-2015, adverse events (AEs) were reported within 5 business days to the Institutional Review Board (IRB) via an AE form and included on the AE log on the annual continuing review application to comply with IRB policy.
Groups:
- No Drug: Tetraplegia: Lesion level C3-T1, ASIA levels A and B, ages 18-68 years
- No Drug: Able-bodied: Age- and gender-matched to individuals with tetraplegia.
- Drug: Tetraplegia: Those individuals with tetraplegia who completed visit 1 of testing (i.e. no drug)
Arm/Group | No Drug: Tetraplegia | No Drug: Able-bodied | Drug: Tetraplegia
Serious Adverse Events (participants affected / at risk) | 1/17 | 0/13 | 1/11
Other Adverse Events (participants affected / at risk) | 1/17 | 0/13 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Drug: Tetraplegia (N=17) | No Drug: Able-bodied (N=13) | Drug: Tetraplegia (N=11)
Autonomic Dysreflexia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) — Subject experienced autonomic dysreflexia (i.e. increased blood pressure, decreased heart rate, diaphoresis) due to a need to be catheterized. Once catheterized, subject's blood pressure and heart rate returned to normal.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Drug: Tetraplegia (N=17) | No Drug: Able-bodied (N=13) | Drug: Tetraplegia (N=11)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Subject experienced neck pain due to excessive muscle tightness, secondary to cold exposure.

LIMITATIONS AND CAVEATS:
Did not assess cognitive performance a third time, after Tcore in the group with tetraplegia had returned to baseline levels.

Study had a small sample size, and only included males.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes